CLINICAL TRIAL: NCT03934892
Title: Prognostic Value of Peak Lactate During Cardiopulmonary Bypass in Adult Cardiac Surgeries: a Cohort Study
Brief Title: Prognostic Value of Peak Lactate During Cardiopulmonary Bypass in Adult Cardiac Surgeries
Status: Completed | Type: Observational
Sponsor: Hualien Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Tso Cheng, Director, Hualien Tzu Chi General Hospital
Other Study IDs: HualienTCGH
Record Dates: First submitted 2019-04-24; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Cardiopulmonary Bypass; Lactate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lactate during CPB: check lactate levels routinely during cardiac operations with cardiopulmonary bypass, choose the peak lactate data
  Interventions: Diagnostic Test: serum lactate

INTERVENTIONS:
Diagnostic Test: serum lactate — check lactate levels during cardiopulmonary bypass in adult cardiac operations

SUMMARY:
Tissue hypoperfusion during cardiopulmonary bypass (CPB) affects cardiac surgical outcomes. Lactate, an end product of anaerobic glycolysis from oxygen deficit, is an obtainable marker of tissue hypoxia. The investigators aimed to determine the value of blood lactate level during CPB in adult cardiac surgeries in predicting outcomes.

The investigators retrospectively reviewed the patients underwent cardiac surgeries with CPB from January 2015 to December 2015. The patient's characteristics, pre-operative status, surgical type, and intra-operative lactate levels were collected. The outcomes were in-hospital mortality and complications. Receiver operating characteristics (ROC) curves were used to assess the ability of peak lactate level during CPB to predict in-hospital mortality.

DETAILED DESCRIPTION:
The baseline characteristics, including age, gender, body mass index (BMI), comorbidities, left ventricular ejection fraction (LVEF, %), European system for cardiac operative risk evaluation II (EuroSCORE II), pre-operative hematocrit, and serum creatinine levels were recorded. The surgical type was classified as coronary artery bypass grafting (CABG), valve surgery, combined surgery including CABG and valve surgery, great vessel surgery including aortic dissection, and other surgeries. The priority of surgery was classified as elective, urgent, and emergent. The intra-operative variables included CPB time, aortic cross-clamp time, initial lactate level at the beginning of the operation, and the peak lactate level during CPB.

ELIGIBILITY:
Inclusion Criteria:

* adults patients underwent cardiac surgeries with cardiopulmonary bypass from January 2015 to December 2015

Exclusion Criteria:

* patients with missing data from records

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults patients underwent cardiac surgeries with cardiopulmonary bypass from January 2015 to December 2015
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | From date of inclusion until date of death from any cause during hospitalization, assessed up to one year
  peak lactate level during cardiopulmonary bypass predicts in-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Yi-tso Cheng, MD, Study Chair — Hualien Tzu Chi General Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD) will be available on request.

REFERENCES:
- [Result] Demers P, Elkouri S, Martineau R, Couturier A, Cartier R. Outcome with high blood lactate levels during cardiopulmonary bypass in adult cardiac operation. Ann Thorac Surg. 2000 Dec;70(6):2082-6. doi: 10.1016/s0003-4975(00)02160-3. PMID 11156124
- [Result] O'Connor E, Fraser JF. The interpretation of perioperative lactate abnormalities in patients undergoing cardiac surgery. Anaesth Intensive Care. 2012 Jul;40(4):598-603. doi: 10.1177/0310057X1204000404. PMID 22813486